CLINICAL TRIAL: NCT05301374
Title: The Effect of Cartoon Watching on Anxiety and Pain During Central Venous Catheter Dressing Changes in Children With Cancer: A Randomized Controlled Trial
Brief Title: The Effect of Cartoon Watching During Central Venous Catheter Dressing Changes in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Pınar BEKAR, Assistant Professor, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAEK-610
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Pain; Anxiety
Keywords: Anxiety; Cancer; Cartoon; Central Venous Catheter; Child; Pain
MeSH Terms: conditions — Pain; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cartoon Group (Experimental): Children in the cartoon group before the procedure, they chose one of the cartoons predetermined by the researchers. The children in the cartoon group started watching a cartoon of their choice 2 minutes before the procedure and they kept watching until the procedure was ended. Parent was with their children during the procedure in both groups.
  Interventions: Behavioral: Watching Cartoon
- Control Group (No Intervention): No intervention was performed to reduce anxiety and pain for children in the control group. Parent was with their children during the procedure in both groups.

INTERVENTIONS:
Behavioral: Watching Cartoon — Children in the cartoon group before the procedure, they chose one of the cartoons predetermined by the researchers. The children in the cartoon group started watching a cartoon of their choice 2 minutes before the procedure and they kept watching until the procedure was ended.
  Arms: Cartoon Group

SUMMARY:
Many medical interventions, including dressing change of central venous catheters, can cause anxiety and pain in children with cancer. The aim of this study is to determine the effect of cartoon watching technique on anxiety and pain during central venous catheter dressing changes in children with cancer.

DETAILED DESCRIPTION:
This was a parallel randomized controlled trial with 80 children with cancer. They were randomly assigned to one of two groups, including 40 children in the control group and 40 children in the cartoon group.

Each child's anxiety was evaluated by the child using the Children's Fear Scale before, during and after central venous catheter dressing changes, and each child's pain during and after the procedure was evaluated by the child using the Wong-Baker Faces Pain Rating Scale. Each child's heart rate and oxygen saturation were measured with a pulse oximeter device before, during and after the procedure.

The children in the cartoon group started watching a cartoon of their choice 2 minutes before the procedure and they kept watching until the procedure was ended.

No intervention was performed to reduce anxiety and pain for children in the control group.

Parent was with their children during the procedure in both groups.

ELIGIBILITY:
Inclusion Criteria:

* 5-12 years old
* a cancer diagnosis
* having a central venous catheter
* not having taken any analgesics in the 6 hours before the procedure
* not having any visual or auditory problems that prevent watching cartoons
* being suitable motor development and cognitive level for watching cartoons
* being a child and parent volunteering to participate in the study
* the absence of any health problems that prevent communication in the parent and the child

Exclusion Criteria:

* the reporting of pain for another reason at the time of the central venous catheter dressing changes
* being of neutropenia
* being in a terminal phase of the disease

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | 4 MONTHS
  Each child's pain during and after the procedure was evaluated with the "Wong Baker Faces Pain Rating Scale" by the child. The scale consists of faces ranging from no hurt (0) to hurts worst (10)

SECONDARY OUTCOMES:
Children's Fear Scale | 4 MONTHS
  Each child's anxiety was evaluated with the "Children's Fear Scale" before, during and after the procedure by the child. It consists of five facial expressions representing a range from no anxiety (0) to severe anxiety (4).
Heart Rate | 4 MONTHS
  The heart rate and oxygen saturation values of the children in both groups were measured and recorded by the researcher before the procedure, during the procedure and after the procedure using a pulse oximeter device.
Oxygen Saturation | 4 MONTHS
  The heart rate and oxygen saturation values of the children in both groups were measured and recorded by the researcher before the procedure, during the procedure and after the procedure using a pulse oximeter device.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Prof.Dr., Study Director — Akdeniz University, Department of Child Health and Disease Nursing
Locations (1):
- Pınar BEKAR, Burdur, Turkey (Türkiye)